CLINICAL TRIAL: NCT00538941
Title: Effects of Swiss Dark Chocolate on Endothelial and Baroreceptor Function and Markers of Inflammation in Patients With Chronic Heart Failure
Brief Title: Effects of Chocolate in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: PD Dr. med. Roberto Corti, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK1124_Chocolate_CHF
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Heart Failure
Keywords: chocolate,; heart failure,; endothelial function,; platelet adhesion,; oxidative stress,; baroreceptor function,
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): daily intake of 40gr chocolate (Nestlé Noir intense) in the morning and 40gr chocolate in the evening.
  Interventions: Dietary Supplement: Nestlé Noir intense 40 grx2
- 2 (Placebo Comparator): Nestlé Placebo Chocolate 40gr in the morning and 40gr chocolate in the evening.
  Interventions: Dietary Supplement: Nestlé Placebo Chocolate 40 grx2

INTERVENTIONS:
Dietary Supplement: Nestlé Noir intense 40 grx2 — daily intake of 40gr chocolate (Nestlé Noir intense or Nestlé Placebo Chocolate) in the morning and 40gr chocolate in the evening.
  Arms: 1
Dietary Supplement: Nestlé Placebo Chocolate 40 grx2 — Nestlé Placebo Chocolate 40 gr in the morning and 40gr chocolate in the evening.
  Arms: 2

SUMMARY:
The aim of the present study is to investigate whether in patients with chronic heart failure endothelial dysfunction and baroreceptor function is altered by ingestion of a flavonoid-rich dark chocolate in comparison to placebo chocolate (Nestlé Placebo Chocolate) on top of standard medication.

Moreover, we will evaluate the effect of chocolate on oxidative stress, platelet adhesion as well as systemic inflammatory response such as C-reactive protein and pro-inflammatory cytokines in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Heart failure ( NYHA ≥II, LVEF<50%, independent of aetiology)
2. Nonsmokers
3. Age: 30-80
4. Written obtained informed consent

Exclusion Criteria:

1. Decompensated Heart failure
2. Instable Angina pectoris
3. Smokers
4. Ventricular tachyarrhythmias or AV-Block >I°
5. Renal failure (>200 umol)
6. Liver disease (ALT or AST >150 IU)
7. Diabetes mellitus
8. Obesity (BMI >30 kg/m2)
9. Symptomatic hypotension, hypertension >160/100mmHg
10. Known allergy to compounds of Nestlé noir intense
11. History of gastric ulcer or bleeding, current diarrhea
12. Venous thrombosis or pulmonary embolism, at present or recurrent history of Infectious disease, acutely or chronic
13. Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
14. Neoplasia (unless healed or remission >5 years)
15. Participation in another study within the last month
16. Concomitant vitamin supplements

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
endothelial function | acute (2 hours), chronic (2 and 4 weeks)

SECONDARY OUTCOMES:
shear-stress dependent platelet function; Oxidative stress; baroreceptor function Systemic inflammatory response (assessed as change in high sensitivity CRP, 8-Isoprostanes, CD-40 ligand); Plasma epicatechins. | acute (2 hours), chronic (2 and 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Noll, MD, Principal Investigator — Cardiovascular Center, University Hospital Zurich, Zurich, Switzerland
Locations (1):
- Cardiovascular Center, Cardiology, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Flammer AJ, Sudano I, Wolfrum M, Thomas R, Enseleit F, Periat D, Kaiser P, Hirt A, Hermann M, Serafini M, Leveques A, Luscher TF, Ruschitzka F, Noll G, Corti R. Cardiovascular effects of flavanol-rich chocolate in patients with heart failure. Eur Heart J. 2012 Sep;33(17):2172-80. doi: 10.1093/eurheartj/ehr448. Epub 2011 Dec 15. PMID 22173910